CLINICAL TRIAL: NCT05124964
Title: Prospective Study on Quality of Life in Patients With Intracranial Germ Cell Tumors
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Tao Jiang, President, Beijing Tiantan Hospital
Other Study IDs: CHN-IGCT-002
Record Dates: First submitted 2021-10-13; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Quality of Life
Keywords: intracranial germ cell tumors; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients with newly diagnosed primary intracranial germ cell tumors are scheduled for subsequent anti-tumor therapy.
  Interventions: Other: PedsQL 4.0 Scale; Other: Short Form-36; Other: Chinese Wechsler Intelligence Scale for Children

INTERVENTIONS:
Other: PedsQL 4.0 Scale — The PedsQL 4.0 Generic Core Scale contains 23 items that measures physical (eight items), emotional (five items), social (five items), and school (five items) functions. The Scale comprises parallel patient self-report and parent proxy-report formats. The items are reverse-scored and trans- formed to a 0-100 scale according to the instructions, and higher scores indicate a better HRQOL. PedsQL 4.0 will be evaluated at baseline, yearly through 3 years post-enrollment.
  Other Names: PedsQL 4.0 Generic Core Scale
Other: Short Form-36 — Altogether, 36 questions with standardized response choices were organized into eight scales, including physical functioning (PF), role limitations as a result of physical health problems (RP), body pain (BP), general health perceptions (GH), vitality (VT), social functioning (SF), role limitations as a result of emotional problems (RE), and general mental health (MH). Additionally, reported health transition (HT) was used to evaluate general health changes during the previous year. The raw scores were converted to a 0-100 scale according to the instructions, and higher scores indicated a better HRQOL. Physical component score (PCS) and mental component score (MCS) were also calculated. SF-36 will be evaluated at baseline, yearly through 3 years post-enrollment.
  Other Names: SF-36
Other: Chinese Wechsler Intelligence Scale for Children — The intelligence of the child was tested by the China-Wechsler Intelligence Scale for Children (C-WISC), which was revised by Gong and Cai at Hunan Medical University. The C-WISC consists of 11 individual tests that include six verbal tests [Information (I), Comprehend (C), Sorting (S), Arithmetic (A), Vocabulary (V), and Digit symbol (D)] and five performance tests [Picture Completing (PC), Picture Arrangement (PA), Block Pattern (BP), Object Assembly (OA), and Coding (CD)]. Based on individual testing, vocabulary scores (V), procedure scores (P), and full scores (F) were obtained. Furthermore, the VIQ, PIQ, and full intelligence quotient (FIQ) were calculated progressively . C-WISC will be evaluated at baseline, yearly through 3 years post-enrollment.
  Other Names: C-WISC

SUMMARY:
The primary purpose of this study is to characterize the quality of life in patients with intracranial germ cell tumors. Those findings can contribute towards a better understanding of the impact of the current treatment strategy on survivors.

DETAILED DESCRIPTION:
The characteristics of the quality of life in patients with intracranial germ cell tumors are far from understood. The main reason is the rare occurrence of the disease. As a result, most findings came from retrospective studies in which only dozens of patients participated. Generally, patients with intracranial germ cell tumors have a good prognosis, especially those with germinoma.

Over 90% of patients with germinoma will survival after ten years of follow-up. Thus, the quality of life in long-term survivors is of concern. The investigators designed this prospective study to address this issue to understand better the characteristics of the quality of life in patients with intracranial germ cell tumors and provide information for optimizing the current treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* 3 years ≤ age ≤ 21 years
* Newly diagnosed primary intracranial germ cell tumors
* Written informed consent

Exclusion Criteria:

* Relapsed disease
* Poor compliance

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with newly diagnosed primary intracranial germ cell tumors are eligible for the study, including those diagnosed based on serum/cerebral spinal fluid tumor marker(s) elevation (β-HCG and/or AFP) and/or pathology.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change of score of the QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales, Chinese edition) | Evaluation will be evaluated at baseline, yearly through 3 years post-enrolment.
  The PedsQL 4.0 Generic Core Scale contains 23 items that measures physical (eight items), emotional (five items), social (five items), and school (five items) functions. The Scale comprises parallel patient self-report and parent proxy-report formats. The items are reverse-scored and trans- formed to a 0-100 scale according to the instructions, and higher scores indicate a better HRQOL. (age ≤18 years)

SECONDARY OUTCOMES:
Change of score of the QoL questionnaire (Short form-36) | Evaluation will be evaluated at baseline, yearly through 3 years post-enrolment.
  Altogether, 36 questions with standardized response choices were organized into eight scales, including physical functioning (PF), role limitations as a result of physical health problems (RP), body pain (BP), general health perceptions (GH), vitality (VT), social functioning (SF), role limitations as a result of emotional problems (RE), and general mental health (MH). Additionally, reported health transition (HT) was used to evaluate general health changes during the previous year. The raw scores were converted to a 0-100 scale according to the instructions, and higher scores indicated a better HRQOL. Physical component score (PCS) and mental component score (MCS) were also calculated. (Age >15 years)

OTHER OUTCOMES:
Change of score of Chinese Wechsler Intelligence Scale for Children | Evaluation will be evaluated at baseline, yearly through 3 years post-enrolment.
  The intelligence of the child was tested by the China-Wechsler Intelligence Scale for Children (C-WISC), which was revised by Gong and Cai at Hunan Medical University. The C-WISC consists of 11 individual tests that include six verbal tests [Information (I), Comprehend (C), Sorting (S), Arithmetic (A), Vocabulary (V), and Digit symbol (D)] and five performance tests [Picture Completing (PC), Picture Arrangement (PA), Block Pattern (BP), Object Assembly (OA), and Coding (CD)]. Based on individual testing, vocabulary scores (V), procedure scores (P), and full scores (F) were obtained. Furthermore, the VIQ, PIQ, and full intelligence quotient (FIQ) were calculated progressively .

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China